CLINICAL TRIAL: NCT03795259
Title: Effect of Rocuronium and Sugammadex Under Sevoflurane and Desflurane Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: GAMZE PİRİNÇ ŞAŞIOĞLU (Unknown); GÜNER KAYA (Unknown); Ayse Cigdem Tutuncu (Other)
Responsible Party: Principal Investigator, pinar kendigelen, MD, Principal investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 83045809-604.01
Record Dates: First submitted 2018-12-27; First posted 2019-01-07 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Anesthetics, Inhalation; Neuromuscular Blockade; Anesthesia, General
Keywords: Sugammadex; Sevoflurane; Desflurane; Rocuronium; TOF; Child; Train-of-four
MeSH Terms: conditions — Respiratory Aspiration | interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Active Comparator): Anesthesia will be induced with thiopenthal 5-6 mg/kg and fentanyl 2 mcg/kg. Then rocuronium 0.6 mg/kg will be given by intravenously and patients will be orotracheal intubated when TOF value reaches 0%. Anesthesia will continue with 2% sevoflurane while the patient is ventilated in volume controlled mode (FiO2: 40%, I/E: 1/1.5, PEEP: 5 cmH2O, tidal volume: 8ml/kg). Continuous TOF measurement will continue until the value reaches %25. At this time, sugammadex 2 mg/kg will be given to measure the time for TOF to reach 90%.
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- Desflurane (Active Comparator): Anesthesia will be induced with thiopenthal 5-6 mg/kg and fentanyl 2 mcg/kg. Then rocuronium 0.6 mg/kg will be given by intravenously and patients will be orotracheal intubated when TOF value reaches 0%. Anesthesia will continue with 6% desflurane while the patient is ventilated in volume controlled mode (FiO2: 40%, I/E: 1/1.5, PEEP: 5 cmH2O, tidal volume: 8ml/kg). Continuous TOF measurement will continue until the value reaches %25. At this time, sugammadex 2 mg/kg will be given to measure the time for TOF to reach 90%.
  Interventions: Drug: Rocuronium; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — After induction, rocuronium 0.6 mg/kg will be given by intravenously and patients will be orotracheal intubated when TOF value reaches 0%.
  Other Names: Esmeron, MSD
Drug: Sugammadex — Continuous TOF measurement will continue until the value reaches %25. At this time, sugammadex 2 mg/kg will be given intravenously.
  Other Names: Bridion, MSD

SUMMARY:
Sugammadex is the first selective relaxant binding agent approved to reverse certain non-depolarizing neuromuscular drugs in patients 2 years old and above. Although it has been in use over the last 10 years, more pharmacological studies are needed to understand its overall effects on participants.

As investigators' primary outcome, the investigators aimed to investigate how differently sugammadex reverses neumuscular blockade caused by rocuronium under general anesthesia maintenance with sevoflurane compared with desflurane. Also, to compare the changes in peak airway pressure. As investigators' secondary outcome, the investigators aimed to compare the changes in heart rate and blood pressures after sugammadex injection under sevoflurane and desflurane general anesthesia.

DETAILED DESCRIPTION:
160 participants aged between 2-10 years old and scheduled for lower urinary tract or minor abdominal surgery will be enrolled in the study. Each participant will be assigned sevoflurane (Group S) or desflurane (Group D) anesthesia at enrollment by drawing lots. Parental consent after written and verbal information will be asked on the morning of the surgery.

Participants will be premedicated with midazolam (0.05 mg/kg, Zolamid, Defarma-Turkey) and ketamine (0.1 mg/kg, Ketalar, Pfizer-USA) and brought into operating theater. Routine monitoring will be done with non-invasive blood pressure (every 5 minutes), continuous peripheral oxygen saturation, continuous 3-lead ECG, body temperature and continuous end-tidal carbon dioxide measurements. Participants will be actively warmed to ensure normo-thermia. Train-of-four (TOF) measurements will be performed on the arm without the vascular access.

Anesthesia will be induced with thiopenthal (5-6 mg/kg, Pental, Ulagay-Turkey) and fentanyl (2 mcg/kg, Talinat, VEM-Turkey). After the participant loses consciousness, TOF calibration will be performed and baseline value will be recorded. Then 0.6 mg/kg rocuronium (Myocron, VEM-Turkey) will be given intravenously and serial TOF measurements at 15 seconds intervals will be taken. The time from TOF of 100% to 0% will be recorded as T1. Participant will be orotracheal intubated when the TOF value is 0%. All the patients will be ventilated with Datex Ohmeda S/5 Avance in a volume controlled ventilation mode (air-oxygen mixture, FiO2: 40%, I/E: 1/1.5, PEEP: 5 cmH2O, tidal volume: 8ml/kg). Participant will receive 2% sevoflurane (Sevoran, Abbvie-Italy) or 6% desflurane (Suprane, Baxter-Belgium) according to their groups.

Non-invasive blood pressure, heart rate and peak airway pressure will be recorded at 5 minute intervals after orotracheal intubation. Continuous TOF measurements will be taken until TOF value reaches 25%. Time from TOF of 0% to 25% will be recorded as T2.

When the TOF value is 25%, 2 mg/kg sugammadex (Bridion, MSD-Greece) will be given intravenously and TOF measurements will continue every 15 seconds. The time from sugammadex injection (TOF of 25%) to TOF of 90% will be recorded as T3. Non-invasive blood pressure, heart rate and peak airway pressure will be recorded at the time of sugammadex injection and at 1st, 2nd, 3rd and 10th minutes. Any reactions to sugammadex will be recorded (anaphylaxis, bronchospasm, etc.).

T1, T2 and T3 of Group S and D will be compared. Non-invasive blood pressure, heart rate and peak airway pressure after sugammadex injection at time 0min, 1min, 2min, 3min and 10min will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Lower urinary tract surgery (cystoscopy, examination under general anaesthesia, circumcision etc.) and inguinal hernia surgery expected no to last more than 2 hours
* ASA I-II

Exclusion Criteria:

* Liver and failure
* Upper airway infection
* Asthma
* Exposure to second hand smoke
* Kidney failure
* Obesity (BMI> 30%)
* Rocuronium allergy
* Muscle disease (myasthenia gravis, muscular dystrophies, etc.)
* Calcium channel blocker use
* Patient or family refusal

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Time from TOF of 25% to 90% after 2 mg/kg sugammadex injection | Up to end of surgery
  When the TOF value reaches 25% from 0% after the anesthesia induction, 2 mg/kg sugammadex will be given to reverse neuromuscular blockade. Continuous TOF monitoring will continue every 15 seconds. The time it takes for TOF to reach 90% is the primary outcome.
Time from TOF of 100% to 0% after 0.6 mg/kg rocuronium injection | Up to end of surgery
  After induction of anesthesia a baseline TOF will be recorded (anticipated 100%). 0.6 mg/kg rocuronium will be injected and TOF will be measured every 15 seconds. The time it takes for TOF to reach 0% is the second primary outcome.
Time from TOF of 0% to 25% after orotracheal intubation | Up to end of surgery
  After TOF reaches 0%, orotracheal intubation will be performed. Continuous TOF monitoring will be done every 5 minutes in first 15 minutes and every 15 seconds afterwards. No additional neuromuscular blocking drugs will be given. The time it takes for TOF to reach 25% is the third primary outcome.
Sugammadex effects on respiratory parameters | Up to 10 minutes post-administration of study intervention
  Peak airway pressure observed at and after sugammadex injection at 1st, 2nd, 3rd and 10th minutes.

SECONDARY OUTCOMES:
Sugammadex effects on heart rate | Up to 10 minutes post-administration of study intervention
  Heart rate observed at and after sugammadex injection at 1st, 2nd, 3rd and 10th minutes.
Sugammadex effects on systolic and diastolic blood pressures | Up to 10 minutes post-administration of study intervention
  blood pressures observed at and after sugammadex injection at 1st, 2nd, 3rd and 10th minutes.
Percentage of Participants Experiencing an Adverse Event (AE) after Administration of Study Intervention | Intraoperative and postoperative first 24 hour.
  Observation bronchospasm and anaphylaxis after sugammadex injection

CONTACTS AND LOCATIONS:
Overall Officials: Guner Kaya, Prof., Study Director — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided